CLINICAL TRIAL: NCT05332886
Title: The Effect of Metaverse-Based Healthy Life Program on Risk Reduction of Non-Communicable Diseases in Youth
Brief Title: Metaverse-Based Healthy Life Program for Youth
Acronym: MetaYouth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayşegül İşler Dalgıç (Other)
Collaborators: Horizon (Industry)
Responsible Party: Sponsor-Investigator, Ayşegül İşler Dalgıç, Prof. Dr., Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 123456789
Record Dates: First submitted 2022-03-24; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Health Risk Behaviors; Healthy Lifestyle; Non Communicable Diseases; Health-Related Behavior; Healthy Eating Index; Healthy Nutrition; Physical Inactivity; Stress, Emotional
MeSH Terms: conditions — Health Risk Behaviors; Noncommunicable Diseases; Health Behavior; Sedentary Behavior; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Parallel Desing Active Comparative Group Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, there will be interventions in both groups, as metaverse-based education and activity programme will be given to the MetaHealth Group and digital health education with a mobile application materials will be given to the MobileHealth Group. In both groups, the participants will be aware that an attempt has been made on them, but since they will not know which group they are in, the participant will be blinded. Since the interventions will be managed by the research team, researcher blinding will not be possible. However, the statistician will be blinded. At the end of the research, the groups will be coded as "A" and "B". Statistical analysis will be made by the statistics expert who is blinded to the groups in the project partner company. After the statistical analysis are made and the research report is written, the situations expressed by A and B will be explained to the statistician. In this way, it is planned to control the bias in statistics and reporting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MetaHealth Group (Experimental): It is intervention group that aims to provide youth with healthy lifestyle behaviors by using metaverse technology.
  Interventions: Behavioral: MetaHealth Group
- MobileHealth Group (Active Comparator): It is comparator group that aims to provide youth with healthy lifestyle behaviors by using mobile application materials with digital health education will be given to the MobileHealth Group.
  Interventions: Behavioral: MobileHealth Group

INTERVENTIONS:
Behavioral: MetaHealth Group — Three metaverse rooms will be created via metaverse technology that aims to develop healthy nutrition, physical activity, and psychological resilience skills to reduce the risk of of NCDs in youth.
  Arms: MetaHealth Group
Behavioral: MobileHealth Group — The intervention aims to develop healthy nutrition, physical activity, and psychological resilience skills using mobile application materials to reduce the risk of NCDs in youth.
  Arms: MobileHealth Group

SUMMARY:
This study was planned within the scope of the call titled "Non-communicable diseases risk reduction in adolescence and youth (Global Alliance for Chronic Diseases - GACD)" with identity number HORIZON-HLTH-2022-DISEASE-07-03. The purpose of this project; is to determine the effect of the Metaverse-Based Healthy Life Program to be developed in the project to support youths in decreasing future risks of developing non-communicable diseases (NCDs) and in gaining healthy lifestyle behaviors (HLBs).

DETAILED DESCRIPTION:
The project consists of three phases. Phase 1 Testing the content, quality, reliability, and usability of the "Metaverse-Based Healthy Life Program for Youth" to be developed within the scope of the project Phase 2 Identifying youth at high risk of chronic non-communicable diseases in the research population Phase 3 Evaluating the effect of "Metaverse-Based Healthy Life Program for Youth" implementation on inculcating healthy lifestyle behaviors in youth

ELIGIBILITY:
Inclusion Criteria:

* Being a university student in the project partner countries and not older than 24,
* Having a score of 130 or lower on the HLBS II in the first stage of the research,
* Determining that BMI ≥ 25-34.99 kg/m2 in the first stage of the research and
* Using a smartwatch during the research,
* Accepting to participate in the research voluntarily

Exclusion Criteria:

* Having chronic diseases (asthma, diabetes, heart, kidney failure, hypertension, cancer, etc.)
* Those who have a drug that they use constantly
* Having a psychiatric diagnosis (depression, anxiety, bipolar disorder, schizophrenia, etc.)
* Having a disease that prevents the use of metaverse (vertigo, vision, hearing, etc.)

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behavior Scale II (HLBS II) | The HLBS II score will evaluate at baseline
  The HLBS II consists of 52 items in total and has 6 sub-factors. Sub-factors are spiritual growth, health responsibility, physical activity, nutrition, interpersonal relationships, and stress management. All items on the scale are positive. The rating is in the form of a 4-point Likert. Never (1), sometimes (2), often (3), regularly (4). The lowest score for the whole scale is 52, and the highest score is 208. The Cronbach Alpha reliability coefficient of the scale is 0.94.
Healthy Lifestyle Behavior Scale II (HLBS II) | The HLBS II score will evaluate at third month
  The HLBS II consists of 52 items in total and has 6 sub-factors. Sub-factors are spiritual growth, health responsibility, physical activity, nutrition, interpersonal relationships, and stress management. All items on the scale are positive. The rating is in the form of a 4-point Likert. Never (1), sometimes (2), often (3), regularly (4). The lowest score for the whole scale is 52, and the highest score is 208. The Cronbach Alpha reliability coefficient of the scale is 0.94.
Healthy Lifestyle Behavior Scale II (HLBS II) | The HLBS II score will evaluate at sixth month
  The HLBS II consists of 52 items in total and has 6 sub-factors. Sub-factors are spiritual growth, health responsibility, physical activity, nutrition, interpersonal relationships, and stress management. All items on the scale are positive. The rating is in the form of a 4-point Likert. Never (1), sometimes (2), often (3), regularly (4). The lowest score for the whole scale is 52, and the highest score is 208. The Cronbach Alpha reliability coefficient of the scale is 0.94.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | The IPAQ-SF score will evaluate at baseline
  The IPAQ-SF is a standardized questionnaire prepared to measure the physical activity of people between the ages of 15 and 65. In the survey, there are 7 questions in total in 4 separate sections about the activities that have been done for a minimum of 10 minutes in the last 7 days. The results obtained in the assessment are calculated as metabolic equivalent task (MET) - min/week.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | The IPAQ-SF score will evaluate at third month
  The IPAQ-SF is a standardized questionnaire prepared to measure the physical activity of people between the ages of 15 and 65. In the survey, there are 7 questions in total in 4 separate sections about the activities that have been done for a minimum of 10 minutes in the last 7 days. The results obtained in the assessment are calculated as metabolic equivalent task (MET) - min/week.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | The IPAQ-SF score will evaluate at sixth month
  The IPAQ-SF is a standardized questionnaire prepared to measure the physical activity of people between the ages of 15 and 65. In the survey, there are 7 questions in total in 4 separate sections about the activities that have been done for a minimum of 10 minutes in the last 7 days. The results obtained in the assessment are calculated as metabolic equivalent task (MET) - min/week.
Positive and Negative Affect Schedule (PANAS-SF) | The PANAS-SF score will evaluate at baseline
  The PANAS-SF is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
Positive and Negative Affect Schedule (PANAS-SF) | The PANAS-SF score will evaluate at third month
  The PANAS-SF is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
Positive and Negative Affect Schedule (PANAS-SF) | The PANAS-SF score will evaluate at sixth month
  The PANAS-SF is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül İşler Dalgıç, Professor, Study Director — Akdeniz University
Locations (1):
- Aysegul ISLER DALGIC, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It has been decided not to share data within the scope of the General Data Protection Regulation.